CLINICAL TRIAL: NCT01854346
Title: Genotype and Behavioral Effects of Social Skills Training in Children and Adolescents With High-functioning Autism Spectrum Disorders, a Randomized Controlled Trial (RCT) and Multicenter Study.
Brief Title: Social Skills Group Training ("KONTAKT") for Children and Adolescent With High-functioning Autism Spectrum Disorders
Acronym: KONTAKT-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Child and Adolescent Psychiatry, Stockholm (Industry); Region Stockholm (Other Government); Stiftelsen Sunnerdahls Handikappfond (Other); The Swedish Research Council (Other Government); The Pediatric Research Foundation at Astrid Lindgren Children's Hospital (Other); Majblomman (Unknown)
Responsible Party: Principal Investigator, Sven Bölte, Professor, PhD, head of pediatric neuropsychiatry unit, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KONTAKT
Record Dates: First submitted 2013-04-20; First posted 2013-05-15 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Autism Spectrum Disorder (ASD); Attention Deficit Hyperactivity Disorder (ADHD); Anxiety; Depression
Keywords: Autism spectrum disorder; Social skills training; Group training; Comorbidity; Intervention; Evidence-based
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social skills group training KONTAKT (Experimental): N= 144 participants are offered group training KONTAKT. The intervention includes 12 (brief intervention) and 24 (long intervention) sessions.
  Interventions: Behavioral: Social skills group training, KONTAKT
- Control group (TAU), the usual intervention / treatment (No Intervention): N = 144 participants are received treatment as usual (pharmacological therapy, family therapy, Cognitive behavioral therapy etc).

INTERVENTIONS:
Behavioral: Social skills group training, KONTAKT — KONTAKT is a manual-based social skills group training for children with high functioning autism spectrum disorder (ASD). The program is based on cognitive behavioral therapy (CBT) principles and knowledge of social cognition. The group treatment includes exercises in social skills as well as discussions of social cognition, social interaction, self-reflection and description of themselves and others. The children are training to make contact, to understand and follow social rules, to become aware of themselves and others, to perceive verbal and nonverbal signals in a communication, to develop problem solving skills and coping strategies to manage conflict and to enhance their self-confidence. Intervention includes 12 (brief intervention) and 24 (long intervention) sessions. Each group consists of 4-8 children/adolescents ant two group leaders. The treatment are conducted in cooperation with both parents and teachers.
  Other Names: Social skills training; Social skills group training; KONTAKT
  Arms: Social skills group training KONTAKT

SUMMARY:
This trial investigates the behavioral effects of manualized social skills training (KONTAKT) in children´s and adolescents with high-functioning autism spectrum disorder with psychiatric comorbidity in a RCT, multicenter study. N = 288 are recruited from 10 child and adolescent psychiatric clinics in Stockholm County. The examination of genetic variants as predictors for outcome and a qualitative study of KONTAKT complete the trial.

DETAILED DESCRIPTION:
There are few randomized controlled trials of social skills group training for the Children's and adolescents with high functioning autism spectrum disorders (HFA)(1). The Objective of this trial is to investigate the behavioral effects of the manualized social skills group training KONTAKT (2,3) and the role of genetic variants for training effects.

ELIGIBILITY:
Inclusion criteria:

* Children and adolescent with High-functioning autism (F84.5, F 84.9 according to International Classification of Diseases (ICD-10). Participants have been investigated with the Autism Diagnostic Observation Schedule (ADOS).
* Normal psychometric range of intelligence, intelligence quotient (IQ)> 70 according to Wechsler Intelligence Scale for Children- Fourth Edition (WISC-IV).
* Comorbid diagnosis: ADHD (F90.0 and F98.8), Anxiety Syndrome (F41.1) and depression (F32.9) according to a best estimate clinical assessment.

Exclusion criteria:

Any behavioral disorder not currently allowing meaningful participation in group-based training for ASD, e.g. presence of clinically diagnosed self-injury, conduct disorder (F91), hyperkinetic conduct disorder (F90.1), antisocial personality disorder (F60.2), borderline personality disorder (F60.3) or any form of schizophrenia or related psychotic disorder (F20-F29).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2012-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) | Baseline, 3 months after training and 3 months follow-up
  Parent and teachers report.

SECONDARY OUTCOMES:
Adaptive Behavior Assessment System II (ABAS II) | Baseline, 3 months after training and 3 months follow-up
  Parent and teachers report.
Developmental Disabilities Modification of the Children's Global Assessment Scale (DD-CGAS) | Baseline, 3 months after training and 3 months follow-up
  Experts report.
Clinical Global Impression-Improvement/Severity (CGI) | Baseline, 3 months after training and 3 months follow-up
  Experts report.
Samples With DNA | 2 weeks after the beginning of the treatment
  Genetic material via saliva-kit will be collected.

OTHER OUTCOMES:
Perceived stress Scale (PSS) | Baseline, 3 months after training and 3 months follow-up
  Parent report.
Barn Under Stress (BUS) | Baseline, 3 months after training and 3 months follow-up
  Self report.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Bölte, PhD, Professor, Principal Investigator — Karolinska Institutet, Center of Neurodevelopmental Disorders (KIND)
Locations (1):
- Child & Adolescent Psychiatry Research Center, KIND, Stockholm, Sweden

REFERENCES:
- [Background] Reichow B, Steiner AM, Volkmar F. Social skills groups for people aged 6 to 21 with autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008511. doi: 10.1002/14651858.CD008511.pub2. PMID 22786515
- [Background] 2. Bölte S., Choque-Olsson N., Swedish version, KONTAKT, Social färdighetsträning i grupp med fokus på kommunikation och social interaktion vid autismspektrumtillstånd enligt Frankfurtmodellen. Hogrefe, 2011.
- [Background] Herbrecht E, Poustka F, Birnkammer S, Duketis E, Schlitt S, Schmotzer G, Bolte S. Pilot evaluation of the Frankfurt Social Skills Training for children and adolescents with autism spectrum disorder. Eur Child Adolesc Psychiatry. 2009 Jun;18(6):327-35. doi: 10.1007/s00787-008-0734-4. Epub 2009 Jan 22. PMID 19165532
- [Background] Choque Olsson N, Bolte S. Brief report: "Quick and (not so) dirty" assessment of change in autism: cross-cultural reliability of the Developmental Disabilities CGAS and the OSU autism CGI. J Autism Dev Disord. 2014 Jul;44(7):1773-8. doi: 10.1007/s10803-013-2029-y. PMID 24379174
- [Background] Choque Olsson N, Flygare O, Coco C, Gorling A, Rade A, Chen Q, Lindstedt K, Berggren S, Serlachius E, Jonsson U, Tammimies K, Kjellin L, Bolte S. Social Skills Training for Children and Adolescents With Autism Spectrum Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Jul;56(7):585-592. doi: 10.1016/j.jaac.2017.05.001. Epub 2017 May 10. PMID 28647010
- [Derived] Choque Olsson N, Rautio D, Asztalos J, Stoetzer U, Bolte S. Social skills group training in high-functioning autism: A qualitative responder study. Autism. 2016 Nov;20(8):995-1010. doi: 10.1177/1362361315621885. Epub 2016 Feb 24. PMID 26912485
- See also: Homepage KIND — http://www.ki.se/kind